CLINICAL TRIAL: NCT07040384
Title: Knee Extensors Activation Device Versus Rolled Towel for Early Quadriceps Activation After ACL Reconstruction: Protocol for a Randomized Controlled Trial
Brief Title: KEA vs Towel for Early Quad Activation Post Anterior Cruciate Ligament Reconstruction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jouf University (Other)
Responsible Party: Principal Investigator, Abdulmajeed Alfayyadh, Assistant Professor, Jouf University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Jouf University; Jouf University (Other: Jouf University)
Record Dates: First submitted 2025-06-18; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: ACL Surgery; Quadriceps Strength
Keywords: Anterior cruciate ligament; quadriceps activation; biofeedback; rehabilitation; electromyography; knee; randomized controlled trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KEA Device Group (Experimental): Participants in this arm will perform quadriceps setting exercises using the Knee Extensors Activation (KEA) device. The device includes an inflatable cushion, pressure gauge, and digital repetition counter. Beginning on postoperative Day 1, participants will complete two supervised sessions daily for five days. Each session includes 3 sets of 10 isometric contractions of the quadriceps, with each contraction held for 5 seconds. The KEA device provides real-time visual feedback, encouraging full-effort contractions. A repetition is only counted when the pressure exceeds a preset threshold and returns to baseline, ensuring correct performance. All sessions are supervised by a physiotherapist.
  Interventions: Device: Knee Extensors Activation (KEA) Device
- Towel Group (Active Comparator): Participants in this arm will perform the same quadriceps setting exercises using a conventional rolled towel placed under the knee. This represents the current standard of care. Beginning on postoperative Day 1, participants will complete two supervised sessions daily for five days. Each session consists of 3 sets of 10 isometric quadriceps contractions with 5-second holds. The physiotherapist provides verbal cues and manually counts repetitions. There is no objective feedback or automated monitoring of contraction effort or repetition quality. All other rehabilitation care is consistent between groups.
  Interventions: Other: Conventional Towel-Based Exercise

INTERVENTIONS:
Device: Knee Extensors Activation (KEA) Device — A portable, non-electric device consisting of an inflatable cushion, pressure gauge, and digital counter. It provides objective feedback during isometric quadriceps exercises after ACL reconstruction. The device encourages full contraction by only counting repetitions that exceed a preset pressure threshold and return to baseline.
  Other Names: KEA Device Group
  Arms: KEA Device Group
Other: Conventional Towel-Based Exercise — Standard rehabilitation method using a rolled towel under the knee during quadriceps setting exercises. Patients perform isometric contractions without feedback or objective measurement. Repetitions are manually counted by the physiotherapist.
  Arms: Towel Group

SUMMARY:
The goal of this clinical trial is to learn if a novel Knee Extensors Activation (KEA) device can improve quadriceps muscle activation in adults after anterior cruciate ligament (ACL) reconstruction surgery. The study focuses on adults aged 18-45 years undergoing primary unilateral ACL reconstruction, a population commonly affected by this injury.

The main questions it aims to answer are:

Does using the KEA device lead to greater quadriceps muscle activation (measured via EMG) by postoperative Day 5 compared to standard care using a rolled towel?

Does the KEA device improve early knee function, reduce pain, and decrease fear of movement compared to the towel method?

Researchers will compare participants using the KEA device versus a control group using the conventional rolled towel during early postoperative rehabilitation to see if the KEA device provides better outcomes.

Participants will:

Begin quadriceps strengthening exercises on the first day after ACL surgery.

Be randomly assigned to use either the KEA device or a rolled towel for isometric quadriceps exercises.

Perform 3 sets of 10 repetitions of knee extension exercises, twice daily for 5 consecutive days.

Undergo assessment of quadriceps EMG activation and complete questionnaires (KOOS, IKDC, TSK, and VAS) on Day 5.

DETAILED DESCRIPTION:
BACKGROUND Rupture of the anterior cruciate ligament (ACL) and its surgical reconstruction are followed by substantial deficits in quadriceps muscle function. In the early postoperative period, reflexive inhibition of the quadriceps, known as arthrogenic muscle inhibition (AMI), leads to drastically reduced voluntary muscle activation. Quadriceps activation failure contributes to weakness, which is concerning since quadriceps strength is strongly related to knee function and stability. Without effective intervention, patients can experience persistent strength deficits, delayed functional recovery, and even altered knee biomechanics due to inadequate quadriceps activation. Notably, one study reported that by 2 weeks after ACL reconstruction, the electromyographic (EMG) activation amplitude of the vastus medialis was less than 50% of normal levels, highlighting the severity of early postoperative quadriceps inhibition.

Early rehabilitation therefore prioritizes reactivation of the quadriceps. Standard ACL rehabilitation protocols universally include quadriceps setting exercises beginning immediately after surgery. Quadriceps setting is an isometric contraction of the knee extensors (quadriceps) with the knee in extension, often performed with a rolled towel or bolster placed under the knee to provide a slight knee flexion angle and a target to press down against. This simple exercise is aimed at recruiting the quadriceps muscle and counteracting AMI as soon as possible. Clinical guidelines and expert consensus recommend initiating such isometric quadriceps contractions on post-op day 1 to restore active knee extension and prevent loss of motion. The conventional method using a rolled towel under the knee is easy and requires no special equipment; however, it provides minimal feedback to the patient. The patient or therapist typically counts repetitions, and the assessment of contraction quality (e.g. how hard the muscle is engaging) is largely subjective.

Enhancing feedback during early exercises may improve quadriceps muscle recruitment. Prior studies have shown that adjunctive biofeedback modalities can significantly improve quadriceps activation and outcomes in early ACL rehabilitation. For example, it's demonstrated that adding electromyographic biofeedback (visual EMG signal feedback) to standard exercises in the first weeks after ACL reconstruction led to greater quadriceps EMG output and better knee extension range than exercise alone. Similarly, neuromuscular electrical stimulation (NMES) is often used alongside exercise to help activate the quadriceps, with evidence that combined NMES and exercise yields stronger quadriceps than exercise alone in the early phase post-ACL. These findings underscore the importance of maximizing muscle activation through innovative rehabilitation strategies during the vulnerable immediate postoperative period.

The Knee Extensors Activation (KEA) Device was developed to address the need for objective feedback and standardization in early quadriceps rehabilitation. The KEA device is a novel, portable tool consisting of an inflatable cushion, a hand-held air pump, an integrated pressure gauge, and a digital repetition counter. The inflatable cushion (placed under the patient's knee) provides resistance during isometric contraction, similar to a rolled towel but with adjustable pressure. The built-in pressure gauge displays the pressure inside the cushion, and is equipped with sensor markers that indicate when a full contraction (sufficient pressure threshold) is achieved. When the patient contracts the quadriceps and presses the knee down on the cushion, a pressure indicator moves; reaching the end-range sensor triggers the digital counter to register a successful repetition. The counter only increments when the pressure has risen above a preset threshold (indicating an adequate contraction) and then returns to baseline, ensuring that only correct, full-effort repetitions are counted. By providing visual feedback of pressure and an automatic rep count, the device aims to engage the patient and encourage maximal activation of the quadriceps with each contraction. In doing so, it standardizes the quad set exercise and reduces reliance on the therapist's subjective judgment of effort or on the patient's inconsistent self-monitoring.

It's hypothesized that using the KEA device in the first week after ACL reconstruction will result in greater quadriceps muscle activation compared to the conventional rolled towel method. It's further hypothesized that patients using the device will report equal or better early functional outcomes, such as reduced pain and kinesiophobia, due to potentially greater confidence in knee contraction and improved knee extension ability. This paper presents the protocol for a two-arm randomized controlled trial designed to test these hypotheses. The trial's primary objective is to compare the quadriceps muscle EMG amplitude during a maximal contraction on day 5 post-surgery between patients trained with the KEA device versus those performing standard care (towel under knee). Secondary objectives include comparing patient-reported outcomes (knee function, pain, and fear of movement) between the two groups at the end of the intervention. We anticipate that the findings will provide evidence on whether an inexpensive, feedback-enhanced device can improve early ACL rehabilitation outcomes, which could have implications for standard postoperative care.

METHODS/DESIGN Study Design and Setting This study is a single-centre, two-arm randomized controlled trial (RCT) employing parallel groups, conducted at a tertiary-care orthopedic hospital. Participants will be enrolled during their inpatient stay following ACL reconstruction. The study design aligns with SPIRIT guidelines for clinical trial protocols, and reporting will adhere to CONSORT standards. Ethical approval has been bending for review process at the Scientific Research Ethics Committee at Jouf University. All participants will provide informed consent prior to enrollment. Figure 6 illustrates the participant flow from recruitment and eligibility screening through randomization, intervention allocation (KEA device versus rolled towel), and subsequent outcome assessments performed at Day 5 postoperatively.

Participants Inclusion criteria involes Adults aged 18-45 years undergoing primary unilateral ACL reconstruction surgery are eligible for the trial. Participants must be within this age range to capture young to middle-aged adults (who are most commonly affected by ACL injuries) and to ensure a relatively homogeneous activity level. They must be undergoing a primary (first-time) ACL reconstruction on one knee (either autograft or allograft, any surgical technique) and be willing and able to participate in postoperative rehabilitation. All participants are required to provide informed consent and comply with the study procedures for the 5-day inpatient intervention and assessments.

Exclusion criteria covers patients will be excluded if they have any condition that could confound the rehabilitation or outcomes. This includes those undergoing bilateral knee surgery (simultaneous both knees, which would make the rehabilitation protocol and EMG measures incomparable), any significant neuromuscular disorder or cognitive impairment that would interfere with performing the exercises or following instructions, or any history of major lower limb surgery in the past year (aside from the current ACL surgery) that could affect muscle function (e.g. recent fractures or surgeries on the involved leg). Patients with concomitant ligament injuries requiring additional extensive repair (other than minor meniscal trim or minor collateral ligament repair) may also be excluded to maintain a relatively uniform rehabilitation course. Table 1 summarizes the inclusion and exclusion criteria.

Sample size would include a target sample of 40 participants (20 per group) has been set. A priori power analysis was performed based on detecting a difference in quadriceps EMG activation between groups at Day 5. We drew on prior research of early quadriceps facilitation: for example, Christanell et al. reported significantly greater vastus medialis EMG output in an EMG-biofeedback group versus controls at 6 weeks post-ACL,5 even with a total sample of 16 patients. Given that finding, we conservatively anticipate a moderate to large effect size for the difference in EMG amplitude at 5 days using the KEA device. Assuming a between-group difference of approximately 15-20% in normalized EMG amplitude (device vs control) with a standard deviation of ~15% (based on variability observed in similar EMG studies),3 we estimate that 16 participants per group would provide 80% power at α=0.05 (two-tailed) to detect a statistically significant difference. Our chosen sample of 20 per group (~40 total) accounts for potential drop-outs or exclusions. The hospital where the trial is conducted performs a high volume of ACL reconstructions, facilitating recruitment of 40 patients within the planned enrollment period (approximately 6-8 months). Participants will be withdrawn from the study if they cannot complete the intervention due to medical complications or if they request to withdraw; replacements will be recruited until the target sample size is reached.

Randomization: After confirming eligibility and obtaining consent, participants will be randomly assigned to either the KEA Device group or the Towel group in a 1:1 ratio. Randomization will be performed using a computer-generated random sequence with random block sizes (to ensure concealment and balance). Allocation will be concealed in opaque sealed envelopes prepared by an independent researcher not involved in patient recruitment or treatment. On the morning of postoperative Day 1 (the day after surgery), the treating physiotherapist will open the envelope to reveal the group assignment. Due to the nature of the intervention, blinding of participants and treating therapists is not possible, patients will know whether they are using the device or a towel, and therapists must instruct accordingly. However, to minimize bias, the outcome assessor (the physiologist conducting the Day 5 EMG tests and administering questionnaires) will be blinded to group allocation. Participants will be instructed not to reveal which training method they used, and the device or towel will not be present during outcome assessments.

Intervention Protocol Both groups will receive a structured quadriceps exercise protocol starting on Postoperative Day 1 (within ~24 hours after surgery) and continuing through Day 5. This corresponds to the typical inpatient period for post-ACL recovery at our institution (patients are kept for intensive physiotherapy and monitoring during the first 5 days). The intervention consists of two supervised exercise sessions per day (morning and afternoon), for a total of 10 sessions over 5 days. Each session focuses on isometric quadriceps contractions (quadriceps setting exercises), performed as 3 sets of 10 repetitions. For each repetition, the patient is instructed to "tighten your thigh muscle and push the back of your knee down" as hard as possible, hold the contraction for 5 seconds, then relax for 5 seconds before the next repetition. After 10 repetitions, a longer rest of 1 minute is given before starting the next set. This dosage (3×10 reps, 5 s hold) is consistent with common early-phase ACL rehab protocols 6 and is intended to provide sufficient activation stimulus without fatiguing the freshly operated limb excessively. A physiotherapist will supervise all sessions to ensure proper technique and safety.

In this study, the intervention protocol varies primarily in the exercise setup and feedback mechanisms between groups. KEA Device Group participants perform quadriceps setting exercises in a long-sitting position using the patented Knee Extensors Activation (KEA) device. The operated knee rests in approximately 20° flexion over an inflatable cushion secured to a stable 8-shaped base. The cushion is inflated to a comfortable level using a hand pump (Figure 4), allowing pressure adjustment to match the patient's rehabilitation stage. During contraction, the patient presses the knee into the cushion, generating internal pressure that moves a dial indicator on the device's panel-mounted gauge. The gauge has two sensor thresholds-midpoint and end-range-used to assess contraction quality. A digital counter records a repetition only when the pressure reaches the upper sensor and subsequently returns below the midpoint, ensuring a complete contraction-relaxation cycle. This feedback mechanism standardises repetition quality and encourages maximal quadriceps activation (Figures 1-3). During each session, the physiotherapist provides verbal cues, verifies 5-second contraction holds, and monitors progress via the counter. Minimal manual support may be given, but no adjunct devices are used. Between sets, the patient rests and adjusts for comfort. The device is removed post-session. Figure 5 illustrates a typical clinical application of the KEA device.

By contrast, the Towel Group (Control) follows the same exercise protocol, three sets of 10 repetitions with 5-second holds, but uses a rolled towel (10-15 cm diameter) under the knee. The patient is instructed to press the knee down onto the towel while the therapist provides verbal feedback and manually counts repetitions. Unlike the KEA group, there is no objective feedback or automated counting. Repetitions are recorded based on visible effort, even if suboptimal, reflecting standard clinical practice. All other elements-frequency, therapist supervision, positioning, and adjunct treatments (e.g. cryotherapy, mobilisation)-are consistent between groups to isolate the effect of feedback and measurement modality. A summary of the intervention protocol for both groups is presented in Table 2. This table outlines the exercise dosage (frequency, sets, reps), duration, and the distinguishing features (use of KEA device vs towel) Outcome Measures All outcome assessments will be conducted on Day 5 postoperatively, immediately following the final intervention session. This time point was selected to capture the acute effects of the 5-day quadriceps training programme. An experienced assessor, blinded to group allocation, will perform all measurements in a clinical rehabilitation setting. Participants will be familiarised with the procedures to ensure consistent and maximal effort.

The primary outcome is quadriceps activation, quantified by surface electromyography (EMG) amplitude of the rectus femoris, vastus medialis and vastus lateralis. EMG amplitude, a validated proxy for muscle activation, reflects motor unit recruitment during contraction. Testing will be conducted in long sitting with the knee supported by a rolled towel (identical for both groups to avoid bias). Participants will perform three 5-second maximal isometric contractions, with 30 seconds rest between trials. Standard Ag/AgCl electrodes will be placed per SENIAM guidelines, and signals will be sampled at 1000 Hz with a 20-450 Hz band-pass filter. Root-mean-square (RMS) EMG will be computed over a steady 3-second segment, and the highest amplitude from the three trials will be recorded. Data will be normalised to the contralateral leg's Day 5 activation, assuming symmetrical capability; if unreliable, raw values will be analysed with body mass index as a covariate. A composite activation score may be derived from the mean of the three muscles. This measure enables between-group comparison in voluntary muscle activation. Additional qualitative markers such as knee extension capacity and muscle tremor during contraction will be noted. As quadriceps activation failure is known to impair functional recovery, even early improvements in EMG may hold clinical relevance.

Secondary outcomes include knee-specific function, pain and psychological readiness, all assessed on Day 5. The Knee Injury and Osteoarthritis Outcome Score (KOOS) evaluates pain, symptoms, ADL, sport and quality of life (0-100 per subscale), widely used in ACL populations. We expect limited change by Day 5 but will explore pain and symptom subscales for potential group differences. The Tampa Scale of Kinesiophobia (TSK) assesses fear of movement, a known barrier in ACL rehabilitation. The TSK may reflect whether real-time feedback from the KEA device influences early confidence. Since early kinesiophobia can hinder recovery, this measure will help evaluate psychological impact. IKDC Subjective Knee Form, a global measure of knee function (0-100), complements KOOS by capturing symptoms and performance.While some sport-related items may be less applicable at this early stage, IKDC still offers insight into initial recovery. Pain will be measured using a 10 cm Visual Analogue Scale (VAS), capturing both average rest pain and peak pain during exercises. As pain can limit muscle recruitment, group comparisons will determine whether the KEA protocol affects perceived discomfort.

All questionnaires (KOOS, TSK, IKDC and VAS) will be completed on Day 5 before EMG testing to avoid influence from muscular effort. Responses will be collected electronically or on paper. In cases where data cannot be obtained (e.g. due to language or cognitive limitations), these will be recorded as missing, although such participants are generally excluded. Table 3 provides an overview of all outcomes and their respective instruments.

Data Collection and Management Demographic data (age, sex, BMI, activity level, etc.) and surgical details (graft type, any concomitant injuries) will be recorded at baseline from medical records. During the 5-day intervention, therapy logs will document session attendance, any missed reps or issues, and any adverse events (e.g. intense pain, device problems). The digital counter readings from the KEA device group will be noted to verify compliance (each session should have 30 counts if fully completed). In the towel group, therapists will similarly log that 3 sets of 10 were attempted. Any deviations (e.g. patient could only do 2 sets due to fatigue) will be documented.

Outcome data on Day 5 will be recorded on case report forms and then entered into a secure database by a data manager blinded to allocation. EMG data will be stored electronically; the EMG signals will be analyzed offline by a blinded analyst who labels the files by code (so as not to know group). We will average the EMG results from the three quadriceps muscles or analyze them separately depending on distribution; primarily, we expect all three to change in the same direction. The database will be checked for errors and locked after entry. We plan to de-identify and share the dataset underlying the results upon publication, in line with open science practices.

Statistical Analysis All analyses will follow the intention-to-treat principle, including all participants in the groups to which they were randomized, regardless of adherence (as long as outcome data are available). Descriptive statistics will summarize baseline characteristics by group to check for any chance imbalances (though randomization should prevent systematic differences). The primary outcome (quadriceps EMG amplitude, e.g. % of reference) will be compared between the KEA and Towel groups using an independent-samples t-test if the data are approximately normally distributed. If the distribution is skewed or variances unequal, we will use a non-parametric Mann-Whitney U test. A repeated-measures or ANCOVA analysis will also be performed if a baseline measure of activation becomes available (for instance, if we consider the contralateral leg as baseline activation, we could use a paired comparison; however, our primary analysis is the between-group comparison at Day 5). Additionally, the three muscles' EMG values may be analyzed using a multivariate approach (MANOVA) to see if there is a consistent group effect across all heads of the quadriceps.

For secondary outcomes (KOOS subscales, IKDC, TSK, VAS), group comparisons will similarly be made with t-tests or non-parametric equivalents. Given the exploratory nature of secondary outcomes at this early time point, adjustment for multiple comparisons for these outcomes will not be applied, but the findings will be interpreted cautiously. Categorical variables (if any) will be compared with Chi-square or Fisher's exact test.

Effect sizes (Cohen's d or rank-biserial for non-parametric) will be calculated to quantify the magnitude of differences. A subgroup or exploratory analysis may be conducted to see if outcomes differ by gender or by graft type, though the sample is likely too small to draw firm conclusions on subgroups. No interim analyses are planned due to the short intervention and follow-up duration.

Missing data: Minimal missing data is anticipated since the outcome assessment is at day 5 in a controlled setting. If a participant misses the day 5 assessment (e.g. due to early discharge or complication), we will attempt to have them return within 1-2 days for testing. If data remain missing, we will not impute primary outcomes (given short-term, we will likely treat it as missing and only analyze available cases). However, sensitivity analyses using last observation carried forward (not really applicable as no prior measure) or assuming worst-case for missing may be done to ensure results are robust.

Safety and Monitoring The intervention (isometric muscle contractions) is low-risk. All patients are routinely prescribed similar exercises after ACL surgery, so no additional risk from participation is expected beyond standard care. Use of the KEA device does not involve electricity or invasive components, and it has been tested for safety (the cushion pressure used is well below any level that could cause harm; the device is sturdy and stable under the knee). Participants will be monitored for any adverse events such as excessive pain, popping sensations, or swelling increases during exercises. If any participant experiences concerning pain or adverse signs, they will pause exercises and if needed withdraw from the intervention (but still be followed for outcome if possible). A Data Safety Monitoring Officer (an independent senior physiotherapist) will periodically review the log of any adverse events. Given the short timeframe, formal interim analysis for efficacy is not applicable, but safety monitoring is continuous.

All investigators and therapists will maintain protocol adherence, and any protocol modifications will be communicated to the ethics committee and updated in the trial registry.

Discussion Quadriceps weakness and impaired activation continue to present a major challenge during the early stages of ACL rehabilitation.The KEA device introduces a novel solution by delivering real-time feedback and objective monitoring during a foundational exercise, quadriceps setting. To our knowledge, this is the first study to rigorously compare a device-assisted training method with the conventional approach in the immediate postoperative phase. Its randomised controlled design strengthens internal validity by isolating the effect of the feedback mechanism. Both groups follow an identical exercise protocol, enabling direct comparison of EMG amplitude, the primary outcome and mechanistic marker of neuromuscular activation. Measuring EMG on Day 5 allows us to capture early training effects; even modest improvements at this stage could be significant, as conventional rehabilitation often fails to elicit full quadriceps activation weeks after surgery.

If the KEA device enhances EMG activation by Day 5, it may indicate early neuromuscular benefit, possibly translating to better strength recovery and earlier functional milestones. However, a lack of between-group difference would suggest either sufficient efficacy of standard care or that a longer intervention duration is required. The short follow-up period is a limitation, and while the study is not designed to assess long-term outcomes, promising findings would warrant future trials with extended observation to explore whether early gains influence 1-3 month recovery trajectories. Although patients are permited to continue exercises after discharge, the unsupervised nature of post-study activity limits conclusions beyond the controlled 5-day period.

A further consideration is blinding and expectancy bias. The KEA group may benefit from motivational effects linked to the novelty and feedback of the device. While therapist contact are matched across groups, the study is not sham-controlled. Nevertheless, the EMG outcome-being objective and assessor-blinded, mitigates expectancy bias. We acknowledge the KEA group may be partially "trained to the test" due to exposure to biofeedback, but increased EMG implies true physiological activation, not just improved performance.

Another factor influencing generalisability is the protocol's reliance on a 5-day inpatient setting, which may not be feasible in all healthcare systems. However, the KEA device is portable and user-friendly, allowing for potential adaptation to outpatient or home settings with appropriate instruction. The feasibility of such remote protocols merits future exploration.

The inclusion of early patient-reported outcomes such as KOOS, IKDC, TSK and VAS adds valuable insight. For instance, reduced TSK scores in the KEA group may suggest enhanced confidence from observing feedback, potentially mitigating early kinesiophobia. Since fear of re-injury can hinder long-term adherence, this early psychological signal is clinically relevant. Pain responses will be monitored carefully, although both groups perform low-load exercises. Pressure discomfort with the device can be mitigated by adjusting inflation, and pilot testing indicated good tolerance.

Although NMES or cryotherapy are not incorporated, commonly used to reduce AMI, this was intentional to isolate the KEA device's mechanical feedback effect. If proven effective, the device may serve as a low-cost, scalable adjunct or alternative to NMES, especially in low-resource settings. Unlike NMES, the KEA requires active effort, potentially enhancing volitional control and neuromuscular retraining.

In summary, this study targets a critical gap in ACL rehabilitation by evaluating whether a simple feedback-based device can facilitate early quadriceps activation. Demonstrating measurable EMG gains within days could support broader adoption of the KEA device and similar technologies, particularly where traditional methods fall short. Conversely, null results would inform current practice and refine future interventions. Findings will be disseminated through peer-reviewed publication and academic conferences, and shared with clinical teams to guide practice. Informal participant feedback will inform device refinement. If validated, the KEA device could be extended beyond ACL recovery, benefiting early rehabilitation in other knee pathologies such as patellar fractures or joint replacements. Additionally, by standardising effort and enabling objective tracking, it holds promise for improving both clinical outcomes and rehabilitation research design. Ultimately, this study will assess whether integrating a real-time feedback tool into early ACL rehab can enhance recovery beyond traditional methods.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 45 years
* Undergoing primary unilateral anterior cruciate ligament (ACL) reconstruction (any graft type, any surgical technique)
* Able and willing to participate in postoperative rehabilitation
* Able to provide written informed consent
* Able to comply with study procedures and complete the 5-day inpatient exercise program

Exclusion Criteria:

* Bilateral knee surgeries (e.g., simultaneous ACL reconstruction on both knees)
* Significant neuromuscular disorders that may affect rehabilitation or EMG readings
* Cognitive impairment that would interfere with understanding or performing exercises
* History of major lower limb surgery within the past year (excluding the current ACL surgery)
* Concomitant injuries requiring extensive repair (e.g., complex ligament reconstructions beyond minor meniscal or collateral work)
* Any medical condition or postoperative complication that would prevent safe participation in the exercise program

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2026-08-25 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
Quadriceps muscle activation (EMG amplitude) | Postoperative Day 5
  Surface electromyography (EMG) amplitude of the rectus femoris, vastus medialis, and vastus lateralis during maximal voluntary isometric contraction. The outcome will be expressed as the root-mean-square (RMS) amplitude from the best of three trials. Higher values indicate greater muscle activation.

SECONDARY OUTCOMES:
Pain intensity at rest and during exercise (VAS) | Postoperative Day 5
  Pain will be measured using a 10 cm Visual Analogue Scale (VAS), scored from 0 (no pain) to 10 (worst possible pain). Two values will be recorded: average resting pain and peak pain during quadriceps exercises.
Knee function (KOOS) | Postoperative Day 5
  The Knee injury and Osteoarthritis Outcome Score (KOOS) will assess pain, symptoms, activities of daily living (ADL), sport/recreation, and quality of life. Each subscale is scored from 0 (worst) to 100 (best).
Fear of movement (Tampa Scale of Kinesiophobia - TSK) | Postoperative Day 5
  The TSK questionnaire assesses fear of movement or re-injury using 17 items scored from 1 to 4, with higher scores indicating greater kinesiophobia.
Global knee function (IKDC Subjective Knee Form) | Postoperative Day 5
  The International Knee Documentation Committee (IKDC) Subjective Knee Form is a patient-reported outcome measure that evaluates symptoms, function, and ability to participate in sports activities. Scores range from 0 to 100, with higher scores indicating better knee function.

CONTACTS AND LOCATIONS:
Overall Officials: Abdulmajeed Alfayyadh, Principal Investigator — Jouf University

IPD SHARING:
Plan to Share IPD: Yes
Surface electromyography (EMG) amplitude data of the quadriceps muscles (rectus femoris, vastus medialis, vastus lateralis)
  Visual Analogue Scale (VAS) pain scores (rest and during exercise)
  KOOS (Knee Injury and Osteoarthritis Outcome Score) subscale scores
  Tampa Scale of Kinesiophobia (TSK) total scores
  IKDC Subjective Knee Form scores
  Basic de-identified demographic data (age, sex, BMI, surgical details)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: August 25, 2025 to December 1, 2026